CLINICAL TRIAL: NCT05394012
Title: Randomized, Blinded, Positive Control Phase 1a Trial to Evaluate the Safety and Immunogenicity of a SARS-CoV-2 mRNA Chimera Vaccine (RQ3013) in Healthy Adults Aged 18-59 Years
Brief Title: A Phase 1a Trial to Evaluate the Safety and Immunogenicity of a SARS-CoV-2 mRNA Chimera Vaccine Against COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Walvax Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai RNACure Biopharma Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RQ3013-004
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — RQ3013 COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RQ3013 (Experimental)
  Interventions: Biological: RQ3013
- Comirnaty (Active Comparator)
  Interventions: Biological: Comirnaty

INTERVENTIONS:
Biological: RQ3013 — Two doses of 30 μg/0.15 mL at an interval of 28 days, or two doses of 60 μg/0.3 mL at an interval of 28 days
  Arms: RQ3013
Biological: Comirnaty — Two doses of 30 μg/0.3 mL at an interval of 28 days
  Arms: Comirnaty

SUMMARY:
This is a phase Ⅰa, randomized, double-blind, positive control trial in healthy adults, intended to evaluate the safety and immunogenicity profile of RQ3013. The study vaccine is administered IM at upper arm deltoid as a two-dose primary series on day 0, 28.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants 18-59 years, and both males and females should be included;
2. Participants who agree to participate in this clinical trial voluntarily and sign the informed consent form, capable of providing valid identification, understanding and complying with the requirements of the clinical protocol.
3. For female participants of childbearing potential, effective contraception measures should be used within 2 weeks prior to participation in this study and the results of the pregnancy test must be negative. Participants must voluntarily agree to use effective contraceptive measures from the time of signing the informed consent to the end of the study (effective contraceptive measures including oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).
4. Body mass index within range of 18~30 kg/m2

Exclusion Criteria:

1. Abnormal results of laboratory screening tests (exceeding the upper or lower limit of the normal reference range by a factor of 1.2) which was clinically significant judged by clinicians at screening;
2. Abnormal vital signs with clinical significance at screening, with systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, or pulse <50 beats/min or >100 beats/min under conscious state, or axillary temperature ≥ 37.3°C at screening;
3. Known allergy, or history of anaphylaxis, or other serious adverse reactions to study vaccine or its excipients;
4. History of human coronavirus infection/diseases, such as severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS);
5. History of COVID-19, or history of close contact with confirmed/suspected COVID-19 patients, or positive results for either SARS-CoV-2 nucleic acid or antibody tests (IgG and IgM) at screening;
6. Administration of antipyretics or painkillers within 24 hours prior to vaccination;
7. Receipt of any COVID-19 vaccine, live attenuated vaccine within 28 days prior to vaccination, subunit and inactivated vaccine within 14 days prior to vaccination;
8. Blood donation or blood loss (≥450 mL), or receipt of blood or blood-related products, including immunoglobulins, within 3 months prior to vaccination; or any planned blood donation or blood products use during the study period.
9. Participants with the following disease:

   1. Any acute diseases or acute attacks of chronic diseases within 7 days prior to vaccination；
   2. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.；
   3. Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 6 months, with exception of inhaled or topical steroids, or short-term use (≤14 consecutive days) of oral corticosteroids；
   4. Currently suffering from or previously diagnosed with infectious diseases, positive screening results for hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, human immunodeficiency virus antibody；
   5. History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders；
   6. Asplenia, or functional asplenia；
   7. Presence of severe, uncontrollable or hospitalization indicated cardiovascular diseases, diabetes, blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and musculoskeletal diseases, or malignant tumors, except for history of well-controlled chronic diseases, such as diabetes, hypertension, etc.;
   8. Participants who cannot tolerate venepuncture, or have a history of needle or blood phobia;
   9. Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that need continuous anticoagulant usage.
10. Drug or alcohol abuse (alcohol intake ≥ 14 units per week), which in the investigator's opinion, would compromise the participant's safety or compliance with the study procedure;
11. History of a major surgery, per the investigator's judgment, within 12 weeks before enrolment, or not achieving full recovery after surgery, or any planned major surgery during the study;
12. Pregnant or lactating females; males whose partner plans to conceive; males or females who plan to donate sperm or eggs;
13. Having participated or being participating in COVID-19 clinical trials, and those being participating or planning to participate in other clinical trials during the study period;
14. Receipt of any investigational or unlicensed products (drug, vaccine, biological product or device) other than the investigational vaccine within 3 months prior to signing the informed consent form, or plan to use them during the study;
15. Presence of any underlying disease or condition which, in the opinion of the investigator, may place the participant at unacceptable risk, make the participant unable to meet the requirements of the protocol, or interfere with the assessment of vaccine elicited response.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Immediate adverse events (AEs) within 30 minutes after each vaccination, solicited local and systemic AEs for within 14 days and unsolicited AEs within 28 days following each vaccination | within 14 days and 28 days following each vaccination

SECONDARY OUTCOMES:
Serious adverse events (SAEs) and adverse event of special interest (AESI) from first vaccination to 12 months after full immunization | from first vaccination to 12 months after full immunization
Changes of laboratory safety measures at day 4 following each vaccination in comparison to pre-vaccination levels | day 4 following each vaccination in comparison to pre-vaccination levels
Live virus GMT, GMFR and seroconversion rates against Beta and Omicron in serum at pre dose 1, 28 days post dose 1 (pre-dose 2), 14, 28 days post dose 2 | pre dose 1, 28 days post dose 1 (pre-dose 2), 14, 28 days post dose 2
Pseudovirus GMT, GMFR and seroconversion rates against SARS-CoV-2 Beta and Omicron strain in serum at pre dose 1, 28 days post dose 1 (pre-dose 2), 14, 28 days post dose 2 | pre dose 1, 28 days post dose 1 (pre-dose 2), 14, 28 days post dose 2
GMT, GMFR and seroconversion rates of S-Protein Specific IgGs at pre dose 1, 28 days post dose 1 (pre-dose 2), 14, 28 days post dose 2 | pre dose 1, 28 days post dose 1 (pre-dose 2), 14, 28 days post dose 2
Live virus GMT, GMFR and seroconversion rates against Beta and Omicron in serum at month 3, 6, 12 months post dose 2 | 3, 6, 12 months post dose 2
  Live virus GMT, GMFR and seroconversion rates against Beta and Omicron in serum at month 3, 6, 12 months post dose 2
Pseudovirus GMT, GMFR and seroconversion rates against SARS-CoV-2 Beta and Omicron strain at month 3, 6, 12 months post dose 2 | 3, 6, 12 months post dose 2
GMT, GMFR and seroconversion rates of S-Protein Specific IgGs at month 3, 6, 12 months post dose 2 | 3, 6, 12 months post dose 2

OTHER OUTCOMES:
Spike protein specific CD4+, CD8+, CD4+IFN-γ+, CD4+IL-2+, CD4+TNFα+, CD4+IL-4+, CD4+IL-13+, CD8+IFN-γ+, CD8+IL-2+, CD8+TNFα+ cytokine profiling (flow cytometry) at baseline and day 7, 14 after the second dose | at baseline and day 7, 14 after the second dose
Spike protein specific cytokine responses by enzyme-linked immunospot (ELISPOT) assay, IFN-γ, IL-2, IL-4 at baseline and day 7, 14 after the second dose | at baseline and day 7, 14 after the second dose
Spike protein specific T memory cell responses: CD4+ and CD8+ TCM(CCR7+CD45RA-), TEM(CCR7-CD45RA), TEMRA (CCR7-CD45RA+) and TSCM(CCR7+CD45RA+CD95+) at baseline and 28 days, 3, 6 months after the second dose | at baseline and 28 days, 3, 6 months after the second dose

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yuan, Study Director — Walvax Biotechnology Co., Ltd.